CLINICAL TRIAL: NCT03926221
Title: Parent-Adolescent Interpersonal Processes in the Science of Behavior Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21_parent_teen_study; R21HD097819 (NIH)
Record Dates: First submitted 2019-04-04; First posted 2019-04-24 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Sleep Deprivation; Adolescent Behavior
MeSH Terms: conditions — Sleep Deprivation; Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PBC_I plus TranS-C (Experimental): The Parent Behavior Change Intervention (PBC-I) is a behavioral intervention intended to teach parent behavior change techniques to better support their adolescents to improve sleep health behavior. The Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) is comprised of cross-cutting interventions, 'core modules' and 'optional modules'. TranS-C is derived and adapted from our previous disorder-focused research, firmly grounded in basic science and treatment literature.
  Interventions: Behavioral: Parent Behavior Change Intervention (PBC-I) and Transdiagnostic Sleep and Circadian Intervention (TranS-C)

INTERVENTIONS:
Behavioral: Parent Behavior Change Intervention (PBC-I) and Transdiagnostic Sleep and Circadian Intervention (TranS-C) — PBC-I will be administered to the parent and TranS-C will be administered to the teenager. Both interventions are cognitive-behavioral and comprised of six weekly sessions. Parent and teenager sessions will be held in parallel.

SUMMARY:
This study seeks to examine a novel interpersonal target; namely, parent-teen conversations about youth health behavior change. The rationale is that parents have profound impacts on teen risk and vulnerability. Yet parents receive minimal training in the elements of conversations that optimally inspire their children toward engaging in healthy behaviors. A theoretically grounded and reliable taxonomy of behavior change techniques (BCTs) will be used as a basis for scientifically deriving the conversational elements, or micro-mechanisms, that reduce parent-teen conflict and facilitate upward spirals of healthful behavior change. This proposal builds on pilot data from a recently completed NICHD-funded R01 in which a sleep treatment improved sleep and reduced risk on selected outcomes in youth. While sleep-related health behaviors will be the focus of this R21, the research is designed to be relevant to a broad range of health behavior change. As part of an Administrative Supplement to the R21 awarded in Fall, 2019, two changes are made. First, measures of psychophysiology have been added to the Hot Topics Task. Second, an independent sample of teens who are healthy sleepers (n = 20), and their parents, will be tested on the protocol twice, 9 weeks apart. This comparison group is included to control for the passage of time and for completing the protocol twice. They do not receive an intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 10 and 18 and living with a parent or guardian
2. Lowest quartile of the widely used and well-validated Children's Morningness-Eveningness Preferences Scale (CMEP; 27 or lower) and
3. Youth self-reported weekday sleep onset time for the past month later than 10:40 pm for 10- to 13-year- olds; 11:00pm for 14-16 year olds, and later than 11:20 for 17-18 year olds at least 3 nights per week;
4. English language fluency;
5. able and willing to give informed assent;
6. at least one parent/primary caregiver who lives in the same household as the teen for at least 50% of the week must participate in all study sessions.

Exclusion Criteria:

1. An active, progressive physical illness directly related to the onset and course of the sleep disturbance;
2. evidence of sleep apnea, restless legs or periodic limb movements;
3. significantly impairing pervasive developmental disorder;
4. history of substance dependence in the past six months;
5. suicide risk; bipolar disorder or schizophrenia or another current Axis I disorder if there is a significant risk of harm and/or decompensation if treatment of that comorbid condition is delayed as a function of participating in any stage of this study;
6. Participants will not be excluded if medications are stable (> 4 weeks).

Inclusion criteria (control group):

1. Age between 10 and 18 and living with a parent or guardian
2. (CMEP; 28 or higher) on Children's Morningness-Eveningness Preferences Scale
3. Item #6 on the Pittsburgh Sleep Quality Index (PSQI) rated 'fairly' or 'very good'
4. English language fluency;
5. able and willing to give informed assent;
6. at least one parent/primary caregiver who lives in the same household as the teen for at least 50% of the week must participate in all study sessions.

Exclusion Criteria (control group)

1. An active, progressive physical illness directly related to the onset and course of the sleep disturbance;
2. evidence of sleep apnea, restless legs or periodic limb movements;
3. significantly impairing pervasive developmental disorder;
4. history of substance dependence in the past six months;
5. suicide risk; bipolar disorder or schizophrenia or another current Axis I disorder if there is a significant risk of harm and/or decompensation if treatment of that comorbid condition is delayed as a function of participating in any stage of this study;
6. Participants will not be excluded if medications are stable (> 4 weeks).

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Number of BCTs used by parent coded from the Hot Topics Task | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Parent measure.
Parent perception of general conflict between parent and child measured via Conflict Behavior Questionnaire | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Parent measure. 20 items each on a true/false scale. Total score ranges from 0 to 20 and is computed by adding up total score points. Higher scores indicate more general conflict.
Decisional balance proportion | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Measured by Decision Balance Worksheet. Youth measure.
Subjective sleep quality measured via Pittsburgh Sleep Quality Index global score | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. 19 items each on a 4-point scale. Global score ranges from 0 to 21 and is computed by totaling seven component scores. Lower scores indicate healthier sleep quality.

SECONDARY OUTCOMES:
Type of BCTs used by parent coded from the Hot Topics Task | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Parent measure.
Number of negative and positive communication behaviors coded from the Hot Topics Task | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Parent measure.
Youth's perception of general conflict between parent and child measured via Conflict Behavior Questionnaire. | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. 20 items each on a true/false scale. Total score ranges from 0 to 20 and is computed by adding up total score points. Higher scores indicate more general conflict.
Youth self-reported motivation of participating in TranS-C/making sleep behavior changes via the Intrinsic Motivation Questionnaire | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. 18 items on a 7-point Likert scale, with three subscales being used: Interest/Enjoyment, Perceived Competence, and Effort/Importance. Total score ranges from 3 to 21 (1-7 for each subscale score) and is computed by averaging items within each subscale and adding the 3 subscale scores.
Regularity in sleep midpoint across the week measured via daily sleep diary | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure.
Regularity in sleep midpoint across the week measured via actigraphy | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure.
Morningness/eveningness preference measured via Children's Morningness Eveningness Preference Scale | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. 10 items are weighed on either 4- or 5-point scales. Total score ranges from 10 to 43 and is computed by adding up total points. Scores between 10 and 20 indicate eveningness, scores between 28 and 42 indicate morningness, scores between 21 and 27 are categorized as neither.

OTHER OUTCOMES:
Number of BCTs used by parent coded from the End of Treatment Conversation | Change from session 1 to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Parent measure.
Type of BCTs used by parent coded from the End of Treatment Conversation | Change from session 1 to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Parent measure.
Number of negative and positive communication behaviors coded from the End of Treatment Conversation | Change from session 1 to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Parent measure.
Number of conflicts and the mean anger intensity for parent | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Measured via Issues Checklist. Parent measure.
Number of conflicts and the mean anger intensity for youth | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Measured via Issues Checklist. Youth measure.
Youth's subjective Bedtime measured via Daily Sleep Diary | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Self-report of Bedtime in hour : minutes. Bedtime discrepancy between weeknights and weekend nights is calculated. Daily Sleep Diary is obtained over a period of 7 days at pre and post assessment.
Youth's subjective Wakeup Time measured via Daily Sleep Diary | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Self-report of Wakeup Time in hour : minutes. Wakeup Time discrepancy between weeknights and weekend nights is calculated. Daily Sleep Diary is obtained over a period of 7 days at pre and post assessment.
Youth's subjective Sleep Onset Latency (SOL) measured via Daily Sleep Diary | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Self-report of SOL in hour : minutes. SOL discrepancy between weeknights and weekend nights is calculated. Daily Sleep Diary is obtained over a period of 7 days at pre and post assessment.
Youth's subjective Wake After Sleep Onset (WASO) measured via Daily Sleep Diary | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Self-report of WASO in hour : minutes. WASO discrepancy between weeknights and weekend nights is calculated. Daily Sleep Diary is obtained over a period of 7 days at pre and post assessment.
Youth's subjective Number of Awakenings measured via Daily Sleep Diary | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Self-report of Number of Awakenings. Number of Awakenings discrepancy between weeknights and weekend nights is calculated. Daily Sleep Diary is obtained over a period of 7 days at pre and post assessment.
Youth's subjective Time in Bed (TIB) measured via Daily Sleep Diary | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Self-report of TIB in hour : minutes. TIB discrepancy between weeknights and weekend nights is calculated. Daily Sleep Diary is obtained over a period of 7 days at pre and post assessment.
Youth's subjective Naps measured via Daily Sleep Diary | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Self-report of Naps in hour : minutes. Naps discrepancy between weeknights and weekend nights is calculated. Daily Sleep Diary is obtained over a period of 7 days at pre and post assessment.
Youth's subjective Total Sleep Time (TST) deviation score from developmental norms measured via Daily Sleep Diary | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. TST in minutes is computed for weeknights and weekend nights by using self-report of daily Bedtime, Wakeup Time, Sleep Onset Latency (SOL), Wake After Sleep Onset (WASO), Naps. TST discrepancy between weeknights and weekend nights is calculated. TST deviation score from developmental norms is calculated. Daily Sleep Diary is obtained over a period of 7 days at pre and post-assessment.
Youth's subjective Sleep Midpoint measured via Daily Sleep Diary | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Sleep Midpoint in hour : minutes is computed for weeknights and weekend nights by subtracting Waketime from Bedtime and dividing the difference by TST [(bedtime-waketime)/TST]. Sleep Midpoint discrepancy between weeknights and weekend nights is calculated. Daily Sleep Diary is obtained over a period of 7 days at pre and post assessment.
Youth's subjective Total Wake Time measured via Daily Sleep Diary | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youths measure. Total Wake Time in minutes is computed for weeknights and weekend nights by adding up Sleep Onset Latency and Wake After Sleep Onset (WASO). Total Wake Time discrepancy between weeknights and weekend nights is calculated. Daily Sleep Diary is obtained over a period of 7 days at pre and post assessment.
Youth's subjective Sleep Efficacy measured via Daily Sleep Diary | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Sleep Efficacy in minutes is computed for weeknights and weekend nights by dividing Total Sleep Time (TST) by Time in Bed (TIB) times 100 (TST/TIB x 100). Sleep Efficacy discrepancy between weeknights and weekend nights is calculated. Daily Sleep Diary is obtained over a period of 7 days at pre and post assessment.
Youth's objective Bedtime measured via Actigraphy | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Objective method of monitoring Bedtime in hour : minutes. Bedtime discrepancy between weeknights and weekend nights is calculated. Actigraphy is obtained over a period of 7 days at pre and post assessment.
Youth's objective Wakeup Time measured via Actigraphy | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Objective method of monitoring Wakeup Time in hour : minutes. Wakeup Time discrepancy between weeknights and weekend nights is calculated. Actigraphy is obtained over a period of 7 days at pre and post assessment.
Youth's objective Sleep Onset Latency (SOL) measured via Actigraphy | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Objective method of monitoring SOL in hour : minutes. SOL discrepancy between weeknights and weekend nights is calculated. Actigraphy is obtained over a period of 7 days at pre and post assessment.
Youth's objective Wake After Sleep Onset (WASO) measured via Actigraphy | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Objective method of monitoring WASO in hour : minutes. WASO discrepancy between weeknights and weekend nights is calculated. Actigraphy is obtained over a period of 7 days at pre and post assessment.
Youth's objective Number of Awakenings measured via Actigraphy | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Objective method of monitoring Number of Awakenings in hour : minutes. Number of Awakenings discrepancy between weeknights and weekend nights is calculated. Actigraphy is obtained over a period of 7 days at pre and post assessment.
Youth's objective Time in Bed (TIB) measured via Actigraphy | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Objective method of monitoring TIB in hour : minutes. TIB discrepancy between weeknights and weekend nights is calculated. Actigraphy is obtained over a period of 7 days at pre and post assessment.
Youth's objective Naps measured via Actigraphy | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Objective method of monitoring Naps in hour : minutes. Naps discrepancy between weeknights and weekend nights is calculated. Actigraphy is obtained over a period of 7 days at pre and post assessment.
Youth's objective Total Sleep Time (TST) deviation score from developmental norms measured via Actigraphy | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. TST in minutes is computed for weeknights and weekend nights by using Bedtime, Wakeup Time, Sleep Onset Latency (SOL), Wake After Sleep Onset (WASO), Naps. TST discrepancy between weeknights and weekend nights is calculated. TST deviation score from developmental norms is calculated. Actigraphy is obtained over a period of 7 days at pre and post-assessment.
Youth's objective Sleep Midpoint measured via Actigraphy | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Sleep Midpoint in hour : minutes is computed for weeknights and weekend nights by subtracting Waketime from Bedtime and dividing the difference by TST [(bedtime-waketime)/TST]. Sleep Midpoint discrepancy between weeknights and weekend nights is calculated. Actigraphy is obtained over a period of 7 days at pre and post assessment.
Youth's objective Total Wake Time measured via Actigraphy | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Total Wake Time in minutes is computed for weeknights and weekend nights by adding up Sleep Onset Latency and Wake After Sleep Onset (WASO). Total Wake Time discrepancy between weeknights and weekend nights is calculated. Actigraphy is obtained over a period of 7 days at pre and post assessment.
Youth's objective Sleep Efficacy measured via Actigraphy | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Youth measure. Sleep Efficacy in minutes is computed for weeknights and weekend nights by dividing Total Sleep Time (TST) by Time in Bed (TIB) times 100 (TST/TIB x 100). Sleep Efficacy discrepancy between weeknights and weekend nights is calculated. Actigraphy is obtained over a period of 7 days at pre and post assessment.
Parent's perception of coercion in parent-child relationship measured via Parent-Child Coercion Scale | Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment
  Parent measure. 9 items each on a 5-point scale. Total score is computed by adding up total points and dividing them by the number of items completed. Total score ranges from 1 to 5. Higher scores indicate more coercion.
Youth's systolic blood pressure reactivity | Change from pre-treatment to post-treatment, which is an average of 9 weeks after the beginning of treatment. For control group: change from the first interview to the final interview, with 9 weeks spaced apart.
  Youth measure. Blood pressure is measured using an ambulatory blood pressure monitor during the Hot Topic Task. Readings will be averaged during the resting and task periods. Reactivity will be calculated as the change score between the resting and task periods.
Youth's diastolic blood pressure reactivity | Change from pre-treatment to post-treatment, which is an average of 9 weeks after the beginning of treatment. For control group: change from the first interview to the final interview, with 9 weeks spaced apart.
  Youth measure. Blood pressure is measured using an ambulatory blood pressure monitor during the Hot Topic Task. Readings will be averaged during the resting and task periods. Reactivity will be calculated as the change score between the resting and task periods.
Youth's heart rate variability | Change from pre-treatment to post-treatment, which is an average of 9 weeks after the beginning of treatment. For control group: change from the first interview to the final interview, with 9 weeks spaced apart.
  Youth measure. Heart rate variability is measured using an ambulatory electrocardiogram during the Hot Topic Task. HRV will be calculated as the root mean square of successive differences (RMSSD), which is the square root of the mean squared differences between successive beat-to-beat RR intervals.
Parent's systolic blood pressure reactivity | Change from pre-treatment to post-treatment, which is an average of 9 weeks after the beginning of treatment. For control group: change from the first interview to the final interview, with 9 weeks spaced apart.
  Parent measure. Blood pressure is measured using an ambulatory blood pressure monitor during the Hot Topic Task. Readings will be averaged during the resting and task periods. Reactivity will be calculated as the change score between the resting and task periods.
Parent's diastolic blood pressure reactivity | Change from pre-treatment to post-treatment, which is an average of 9 weeks after the beginning of treatment. For control group: change from the first interview to the final interview, with 9 weeks spaced apart.
  Parent measure. Blood pressure is measured using an ambulatory blood pressure monitor during the Hot Topic Task. Readings will be averaged during the resting and task periods. Reactivity will be calculated as the change score between the resting and task periods.
Parent's heart rate variability | Change from pre-treatment to post-treatment, which is an average of 9 weeks after the beginning of treatment. For control group: change from the first interview to the final interview, with 9 weeks spaced apart.
  Parent measure. Heart rate variability is measured using an ambulatory electrocardiogram during the Hot Topic Task. HRV will be calculated as the root mean square of successive differences (RMSSD), which is the square root of the mean squared differences between successive beat-to-beat RR intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Harvey, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No